CLINICAL TRIAL: NCT00267202
Title: A 26-week, Randomized, Double-blind, Parallel-group, Placebo-controlled,Multi-center Study to Evaluate the Effect of Omalizumab on Improving the Tolerability of Specific Immunotherapy in Patients With at Least Moderate Persistent Allergic Asthma Inadequately Controlled With Inhaled Corticosteroids
Brief Title: Study to Evaluate the Effect of Omalizumab on Improving the Tolerability of Specific Immunotherapy in Patients With Persistent Allergic Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Genentech, Inc. (Industry); Tanox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIGE025AUS23
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Results first posted 2011-05-16 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2011-10

CONDITIONS: Allergic Asthma
Keywords: Allergic Asthma, IgE, immunotherapy, omalizumab
MeSH Terms: conditions — Epilepsy, Idiopathic Generalized | interventions — Omalizumab; Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): The dose of placebo was determined according to the omalizumab US product label using a dosing table nomogram that ensures patients receive at least 0.016 mg/kg/IgE (IU/ml) per 4 weeks. The study drug was administered by subcutaneous injection every 2 or 4 weeks according to the dosing table nomogram.
  Interventions: Drug: Placebo; Drug: Immunotherapy
- Omalizumab (Experimental): The dose of omalizumab was determined according to the omalizumab US product label using a dosing table nomogram that ensures patients receive at least 0.016 mg/kg/IgE (IU/ml) per 4 weeks. The study drug was administered by subcutaneous injection every 2 or 4 weeks according to the dosing table nomogram.
  Interventions: Drug: Omalizumab; Drug: Immunotherapy

INTERVENTIONS:
Drug: Placebo — Doses of placebo were administered subcutaneously every 2 to 4 weeks according to the US product label, depending on the patient's body weight and baseline serum IgE.
  Arms: Placebo
Drug: Omalizumab — Doses of omalizumab were administered subcutaneously every 2 to 4 weeks according to the US product label, depending on the patient's body weight and baseline serum IgE.
  Arms: Omalizumab
Drug: Immunotherapy — Customized allergen extracts were prepared centrally for each patient based on his/her specific skin test results. Four vials containing dilutions of the patient's extract were provided. Investigators initiated dosing according to the protocol for the cluster dosing titration regimen, beginning with vial #4 (the most dilute) and progressing to vial #1, which was the most concentrated or "maintenance" solution. Each dose was administered subcutaneously into the deltoid region as a single injection. During study visits that required multiple IT injections, each injection was to be given at least 30 minutes apart. During weeks that required multiple visits for IT injections, each visit was to be separated by at least 48 hours.
  Arms: Placebo
Drug: Immunotherapy — Customized allergen extracts were prepared centrally for each patient based on his/her specific skin test results. Four vials containing dilutions of the patient's extract were provided. Investigators initiated dosing according to the protocol for the cluster dosing titration regimen, beginning with vial #4 (the most dilute) and progressing to vial #1, which was the most concentrated or "maintenance" solution. Each dose was administered subcutaneously into the deltoid region as a single injection. During study visits that required multiple IT injections, each injection was to be given at least 30 minutes apart. During weeks that required multiple visits for IT injections, each visit was to be separated by at least 48 hours.
  Arms: Omalizumab

SUMMARY:
This study is designed to investigate the use of omalizumab as a pretreatment for patients with persistent allergic asthma who are candidates for allergen immunotherapy (ie, allergy shots) and will test the hypothesis that omalizumab may reduce the rate of systemic reactions to immunotherapy in patients with persistent allergic asthma.

ELIGIBILITY:
Inclusion Criteria:

Patients were eligible for inclusion if they met all of the following criteria:

Informed Consent

* Patients who were informed of the study procedures and medications and provided their written informed consent

Demographics

* Male or female
* Any race
* Ages 18 - 55 years
* Body weight >=20 kg and <=150 kg
* Total serum IgE concentration >=30 and <=700 IU/mL at Visit 0

Disease Definitions/Medications

* History of at least moderate persistent allergic asthma (consistent with Global Initiative for Asthma [GINA] guidelines of >=1 year in duration
* On a stable asthma treatment regimen including inhaled corticosteroids for the preceding 4 weeks
* An FEV1 while withholding short-acting beta-agonists for at least 6 hours and long-acting beta-agonists for at least 12 hours, of >=75% of the predicted value at Visit 0
* Evidence of reversible airway obstruction, as defined by an increase in FEV1 of >=12% between 20 to 30 minutes after 4 puffs (or less at the discretion of the investigator) of inhaled short-acting beta-agonist administration at Visit 0 or within the preceding year
* Documented sensitivity to perennial aeroallergens, as evidenced by a positive skin test (wheal >=5mm greater than saline control) to at least 1 of 3 perennial aeroallergens (house dust mite, cat, or dog) at Visit 0 or within the preceding year
* Average PEFR variability <=20% (calculated as [(PM PEF - AM PEF)/(PM PEF + AM PEF)/2 x 100) during the 2-week screening period
* Pre-specified level of nocturnal asthma symptoms (i.e., a mean nocturnal asthma score of >0 and <=0.5) and a mean combined clinical symptom score (nocturnal, morning, and daytime) of >0 and <=3 during the screening period
* Non-smoker for at least 1 year prior to Visit 1, with a smoking history of no more than 10 pack-years (i.e., 1 pack [20 cigarettes] per day for 10 years)
* Judged to be in good physical and mental health (except for his/her asthma), based on medical history, physical examination, and routine laboratory data, and appeared to be able to successfully complete this trial

Exclusion Criteria:

Patients were to be excluded from participation if they met any of the following criteria:

Pulmonary

* History of intubation for asthma
* Asthma exacerbation requiring treatment with systemic steroids within the preceding 3 months
* Asthma exacerbation requiring treatment in an emergency department or a hospital admission in the preceding 6 months
* Upper respiratory tract infection or sinusitis within the preceding 4 weeks
* History of an anaphylactic allergic reaction (except to stinging insects, foods, or drugs other than omalizumab)
* History of treatment with immunotherapy to any allergen within past 3 years
* History of aspirin or non steroidal anti-inflammatory drug (NSAID)-related asthma; patients could have been included in NSAIDs use was avoided for the duration of the study

General Medical

* History of or current malignancy
* Any clinically significant uncontrolled systemic disease or a history of such disease (e.g., infectious, hematologic, renal, hepatic, endocrinologic, gastrointestinal, or cardiovascular disease) within the previous 3 months
* Clinically significant laboratory abnormalities at Visit 1
* Platelet levels <=130 x 10 9/L at visit 1
* Women of childbearing potential who were not practicing a medically approved contraception method (e.g., oral, subcutaneous, mechanical, or surgical contraception), as well as women who were pregnant or nursing
* History of hypersensitivity to any ingredients, including excipients (sucrose, histidine, or polysorbate 20) of the study medication or drugs related to omalizumab (e.g., monoclonal anti-bodies or polyclonal gammaglobulin)
* Severe medical condition(s) that, in the view of the investigator, prohibited participation in the study
* Previous treatment with omalizumab within 1 year of screening
* Considered by the investigator to be potentially unreliable or who may not have reliably attended study visits
* History of drug or alcohol abuse

Procedural

* Unable to perform acceptable, reproducible spirometry, or PEFR measurements
* Unable or unwilling to comply with the study procedures as determined during the screening phase, including adequate completion of the diary

Medications

Patient took the following medications before Visit 0. These medications were not permitted during the trial unless otherwise specified:

* Oral, intravenous, intramuscular, or intra-articular corticosteroids within 4 weeks
* Beta-adrenergic antagonists (including ocular preparations) within 1 week
* Antihistamines within 1 week; after skin testing was completed (Visit 0), antihistamines could be used as needed for the remainder of the study
* Intravenous gammaglobulin or immunosuppressants within 4 weeks
* Tricyclic antidepressants within 1 week
* Investigational drugs within 4 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 275 (Actual)
Dates: Start 2005-12; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- See also: Novartis patient recruitment website — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Omalizumab
Started | 136 | 139
Completed | 83 | 105
Not Completed | 53 | 34
Not completed — Unsatisfactory therapeutic effect | 21 | 8
Not completed — Withdrawal by Subject | 12 | 15
Not completed — Adverse Event | 13 | 7
Not completed — Protocol Violation | 2 | 3
Not completed — Administrative problems | 2 | 1
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Omalizumab | Total
Number analyzed (Participants) | 136 | 139 | 275
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (10.02) | 38.2 (9.89) | 38.2 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 88 | 187
  Male | 37 | 51 | 88
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1
  Black or African American | 11 | 17 | 28
  White | 112 | 118 | 230
  Unknown or Not Reported | 13 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Systemic Allergic Reactions (SAR) to Specific Immunotherapy (SIT)
Description: The number of participants with Systemic Allergic Reactions (SAR) to Specific Immunotherapy (SIT). A SAR was captured and recorded as an outcome, not as adverse events (AEs) or SAEs. The primary analysis time point was the end of Period 4 (maintenance immunotherapy). Participants were observed for 1 hour after each immunotherapy (IT) injection visit. Allergic reactions were graded on a 4-point scale from Grade 1 to Grade 4. Grade 1: Skin symptoms, Grade 2: Gastrointestinal symptoms, Grade 3: Respiratory symptoms and Grade 4: Cardiovascular symptoms.
Time Frame: 26 Weeks
Population: Efficacy Population: Consisted of all randomized patients who completed the omalizumab or placebo treatment period and received at least one dose of immunotherapy.
Measure: Number; unit: participants
Arm/Group | Placebo | Omalizumab | All Patients
Number analyzed (Participants) | 122 | 126 | 248
participants | 32 | 17 | 49

2. Secondary Outcome: Severity of First Systemic Allergic Reaction (SAR)
Description: Systemic reactions associated with immunotherapy (IT), defined as occurring within 1 hour following injection of SIT, were graded on a four-point scale: Grade 1: Skin symptoms (generalized urticaria, itching, or erythema), Grade 2: Gastrointestinal symptoms (stomach pain, nausea, or vomiting), Grade 3: Respiratory symptoms (clinically significant nasal symptoms and/or dyspnea, wheezing, persistent cough, etc.), Grade 4: Cardiovascular symptoms (cyanosis, hypotension, collapse, arrhythmias, or angina pectoris).
Time Frame: 26 Weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Omalizumab | All Patients
Number analyzed (Participants) | 32 | 17 | 49
participants
  Grade 1 (skin symptoms) | 6 | 7 | 13
  Grade 2 (gastrointestinal symptoms) | 0 | 2 | 2
  Grade 3 (respiratory symptoms) | 24 | 6 | 30
  Grade 4 (cardiovascular symptoms) | 2 | 2 | 4
  No systemic allergy | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Who Achieved Target Maintenance Specific Immunotherapy (SIT) Dose
Description: Achievement of target maintenance IT dose is defined as answering 'Yes' to the question, 'Was the target maintenance SIT dose achieved?' on Visit 13, Week 16.
Time Frame: 16 Weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Omalizumab | All Patients
Number analyzed (Participants) | 122 | 126 | 248
participants | 88 | 110 | 198

4. Secondary Outcome: Number of Participants Requiring 8 to 20 Visits to Complete Cluster Specific Immunotherapy (SIT) Dosing Regimen
Description: During period 3, a cluster dosing protocol was utilized to initiate the allergen immunotherapy (IT). Participants received escalating doses of IT according to a cluster dosing titration regimen. Visits 5 through 13 were cluster visits for this study. The number of visits needed for completion of the cluster SIT dosing regimen was defined as the number of planned visits plus the number of unplanned visits needed to reach maintenance IT dose.
Time Frame: Up to 26 Weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Omalizumab | All Patients
Number analyzed (Participants) | 122 | 126 | 248
participants
  8 Visits | 87 | 110 | 197
  9 Visits | 35 | 15 | 50
  10 Visits | 0 | 0 | 0
  11 Visits | 0 | 1 | 1
  12-20 Visits | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Requiring 0 to >=5 Doses of Rescue Medications for Systemic Allergic Reactions (SARs) to Specific Immunotherapy (SIT)
Description: Epinephrine for injection, antihistamines, corticosteroids for injection, inhaled beta-agonists, and oral corticosteroids, as well as other drugs used for managing acute allergic reactions to SIT, were available during all study visits. One dose of rescue medication for SAR reactions was equivalent to 1 entry of the CRF page 'concomitant medications/significant non-drug therapies associated with immunotherapy' in response to the question 'Was this medication given in response to a SAR?'
Time Frame: Up to 26 Weeks
Population: Efficacy population: Consisted of all randomized participants who completed the omalizumab or placebo treatment period, received at least one dose of immunotherapy and received rescue therapy.
Measure: Number; unit: participants
Arm/Group | Placebo | Omalizumab | All Patients
Number analyzed (Participants) | 32 | 17 | 49
participants
  All rescue medications: 0 doses | 2 | 4 | 6
  All rescue medications: 1 dose | 10 | 3 | 13
  All rescue medications: 2 doses | 5 | 3 | 8
  All rescue medications: 3 doses | 4 | 4 | 8
  All rescue medications: 4 doses | 5 | 2 | 7
  All rescue medications: >= 5 doses | 6 | 1 | 7

ADVERSE EVENTS:
Arm/Group | Omalizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 4/139 | 3/136
Other Adverse Events (participants affected / at risk) | 88/139 | 91/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=139) | Placebo (N=136)
Swollen tongue (Gastrointestinal disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sexual abuse (Social circumstances) | 1 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=139) | Placebo (N=136)
Injection site erythema (General disorders) | 20 | 22
Injection site induration (General disorders) | 8 | 8
Injection site pruritus (General disorders) | 19 | 24
Injection site reaction (General disorders) | 28 | 20
Injection site swelling (General disorders) | 14 | 16
Injection site urticaria (General disorders) | 9 | 6
Nasopharyngitis (Infections and infestations) | 16 | 17
Sinusitis (Infections and infestations) | 7 | 13
Upper respiratory tract infection (Infections and infestations) | 19 | 14
Viral upper respiratory tract infection (Infections and infestations) | 3 | 7
Headache (Nervous system disorders) | 7 | 11
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.